CLINICAL TRIAL: NCT06567899
Title: Mechanistic Underpinnings of Preeclampsia
Acronym: MUP
Status: Not yet recruiting | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00004565
Record Dates: First submitted 2024-05-29; First posted 2024-08-23 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood, cord blood, and placenta will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Non-pregnant with previous normal pregnancy: Non pregnant females
- Non-pregnant with previous known preeclampsia: Women with known preeclampsia in previous pregnancy
- First Trimester Pregnant (First antenatal visit): Women in first trimester
- Second Trimester Pregnant: Women in second trimester
- Third Trimester with known preeclampsia: Women in third trimester with diagnosis of preeclampsia
- Third Trimester with Normal Pregnancy: Women in third trimester with no complications.

SUMMARY:
Preeclampsia is a dreadful disease with significant morbidity and mortality. Despite decades of research, we still need a proper diagnostic test or therapeutic option to treat this disorder. The proposed study will determine the diagnostic value of PBMC-secreted sFlt1 and determine the molecular mechanisms involved in its secretion. The molecular mechanisms can be novel therapeutic targets to treat this disorder.

ELIGIBILITY:
Healthy Adults:

• Healthy non-pregnant with previous normal pregnant women

Non-Health Adults:

• Patients will be admitted with the diagnosis of preeclampsia according to the internationally accepted definition of preeclampsia: Blood pressure measurement of 140/90 mm Hg or an increase of 30 mm Hg systolic or 15 mm Hg diastolic over baseline values on at least two occasions, six or more hours apart and proteinuria; 300 mg/24 hour after 20th week of gestation.

Pregnant Women:

Groups 3 - 6 will include pregnant women at different trimesters.

Criteria common to all groups:

* The study will be conducted only in females aged 18 or above.
* Patients in all the groups will be matched for age, which will be 18 or above.
* Women will be matched for body mass index; criteria for normal body mass index will be used based on the Center for Disease Control and Prevention Guidelines.
* Patients with premature rupture of the membrane, non-preeclamptic preterm labor, IUGR, placental abruption, twin? Any other complications during the pregnancy will be excluded from the study.
* Patients with any evidence of genetic or non-genetic malformations of the fetus will be excluded from the study.
* The study will be conducted on women who are non-smokers and do not consume alcohol or recreational drugs.
* The study will be conducted only on primigravida females to minimize phenotyping variability.
* The women with a known history of any chronic disorder, including but not limited to hypertension, diabetes, pulmonary, renal, cardiac, or cerebrovascular disorders, will be excluded from the studies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females and women with desire to get pregnant.
Study Population: Women above 18 years of age.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-07-25 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
sFLT1 levels | Outcome will be measured at 12 weeks, 24 weeks and 36 weeks of pregnancy.
  sFLT1 levels in preeclampsia should be higher than normal pregnancy.

IPD SHARING:
Plan to Share IPD: No